CLINICAL TRIAL: NCT04759430
Title: The Effects of Telerehabilitation and Supervised Stabilization Exercises on Pain, Functionality, Kinesiophobia and Quality of Life in Individuals With Nonspecific Chronic Low Back Pain: A Single Blind Randomized Controlled Trial
Brief Title: The Effects of Telerehabilitation and Supervised Stabilization Exercises in Individuals With Nonspecific Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Ceren Karaduman, Physical Therapist, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1506581
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Low Back Pain
Keywords: chronic pain; exercise; low back pain; quality of life; telerehabilitation
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The individuals are randomly allocated into supervised group, telerehabilitation group and control group
Who Masked: Outcomes Assessor
Masking Description: The researcher who will make the measurements will not know the treatment groups of the individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Group (Active Comparator): 24 individuals will participate in the Supervised group. Patients in the supervised group will be treated individually by the researcher at the hospital. During the application, individuals will apply ten different stabilization exercises in company with a physiotherapist. Exercises will be applied under the supervision of a physiotherapist in the center where the work will be done for 20-30 minutes in each session, three days a week, for a total of 12 sessions for four weeks. The exercises program to be applied to the participants in the group is listed below: Supine position; Abdominal bracing, while continuing the abdominal bracing; heel slides, bridging, 90 degrees hip flexion. Quadruped position; Abdominal bracing while continuing the abdominal bracing; single arm lift, single leg lift, cross-arm leg raises activities. Standing position; Abdominal bracing.
  Interventions: Other: Supervised Group
- Telerehabilitation Group (Experimental): 24 individuals will participate in the Telerehabilitation group. Patients in the telerehabilitation group will attend the treatment from their homes. The exercises will be performed online with the patient by the researcher physiotherapist and supervised through the video conference or phone. The same stabilization exercises will be applied to the participants in the supervised group. Exercises will be applied for 20-30 minutes in each session, three days a week, for a total of 12 sessions for four weeks.
  Interventions: Other: Telerehabilitation group
- Control Group (No Intervention)

INTERVENTIONS:
Other: Supervised Group — Individuals will apply ten different stabilization exercises in company with a physiotherapist.
  Arms: Supervised Group
Other: Telerehabilitation group — Same stabilization exercises will be performed online with the patient by the researcher physiotherapist and supervised through the video conference or phone.
  Arms: Telerehabilitation Group

SUMMARY:
This study aims to investigate the effects of telerehabilitation and supervised stabilization exercises on pain, functionality, kinesophobia and quality of life in individuals with non-specific chronic low back pain. 72 individuals who voluntarily agree to participate in the study will be included. This study divides the patients in three groups: the supervised group: face-to-face stabilization exercises are applied, the telerehabilitation group: treatment through online meetings, and the control group: patients will do home-based exercises that prescribed by physiothrerapist. Evaluations will be made by the same physiotherapist. The researcher who will make the measurements in this study will not know which treatment program was applied to the participants. In this study, The same stabilization exercises will be applied in three different groups. Ten different stabilization exercises will be applied to the participants. Exercises will be performed for 20-30 minutes in each session, three times a week, for four weeks in total, twelve sessions. Clinical and demographic data of the 72 people participating in the study will be taken before treatment. Participants will also fill out questionnaires before and after the treatment that involve; the Oswestry Disability Index to measure(ODI) daily life activity limitations; the Visual Analogue Scale(VAS) for assessing the intensity of pain; Tampa Scale for Kinesiophobia(TSK) to assess fear of movement; and the Short Form(SF-36) in order to assess self-perceived health-related quality of life. Statistical analysis is going to be used in this research through the SPSS 20.0 package program.

DETAILED DESCRIPTION:
Today, low back pain is one of the most common health problems in the world in which create a considerable individual, social and financial burden on the society. Low back pain is classified as specific and nonspecific. While, 10 percent of the paints are suffered from specific low back pain, non-specific low back pain is occured in approximately 90 percent of the population. If low back pain persists for six weeks, it is classified as acute back pain, subacute back pain between six weeks and three months, and chronic low back pain if it lasts for more than three months.

Chronic low back pain (CLBP) is a complex problem that continues for a long time without a cause and is the most common in the musculoskeletal system, leading to disability. Individuals with CLBP have a lower quality of life than the general population. It causes individuals to decrease their activities due to pain and prepares the ground for the continuation of pain. Lack of movement caused by pain in individuals; It negatively affects the quality of life by triggering the continuation of symptoms, causing a decrease in functional levels, limitation in daily life activities, problems in family and work life. There are many physical, psychological and social factors that cause low back pain to become chronic. Age, race, occupation, obesity, smoking, alcohol consumption and stress are the most important factors that trigger the chronicity of low back pain. The effectiveness of a multidisciplinary treatment program and determination of risk factors in the management of CLBP is known. Treatment approaches include medical treatment, surgical treatment and physiotherapy applications. In physiotherapy programs, patient education, back schools, electrotherapy applications, traction, massage, superficial heat applications, corsets and exercise approaches are used. Stretching exercises, trunk flexion-extension exercises, resistantce exercises, stabilization exercises are the main exercise approaches used to cope with low back pain. In addition to exercises performed under the supervision of a physiotherapist, home exercise programs are also provided for low back pain. Stabilization exercises have various benefits on the musculoskeletal system. Stabilization exercises that aim to protect and support the spine by regenerating muscle control, applied in muscle activation losses caused by injury or degenerative changes, increase strength and flexibility. Stabilization exercise has been reported to be effective in reducing pain and improving functional disability in patients with nonspecific CLBP, improving individuals psychologically and also increasing the quality of life of patients. Stabilization exercises have been found to be effective in increasing the cross-sectional area of the lumbar multifidus muscle, which is one of the muscles needed to maintain the proper stability of the spine.

Today, in line with technological developments, the use of common information processing, sensor networks, three-dimensional (3D) computer graphics, internet and mobile phone applications in healthcare services is widespread. Telerehabilitation refers to the provision of rehabilitation services through information and communication technologies. Clinically this term; covers a range of rehabilitation and habilitation services including assessment, monitoring, prevention, response, control, training, consultation and counseling. Along with telerehabilitation, rehabilitation practices can be applied in health centers as well as homes, schools or community-based work sites. Mostly, there are studies in the literature regarding its use in musculoskeletal disorders, coronary heart disease, some types of cancer, type 2 diabetes, hypertension and physically disabled individuals. Due to the social distance and isolation, which are the effects of the covid-19, which spread in a short time in our country and all over the world, there are disruptions in individuals' continuing their treatment. Telerehabilitation allows one-to-one physiotherapist-patient meetings without the need for contact and provides flexibility to patients in terms of time. Exercise is one of the treatments that physiotherapists can give using telerehabilitation. With the applications made with telerehabilitation, individuals are provided to take an active role in their own rehabilitation and individuals can have the ability to manage themselves.

ELIGIBILITY:
Inclusion Criteria:

* Having non-specific chronic low back pain
* Non-specific chronic low back pain ⩾three months
* Being over the age of 18
* Score of ⩾4 on the Roland-Morris Disability Questionnaire (RMQ)
* Agree to voluntarily participate in the research

Exclusion Criteria:

* Presence of lumbar stenosis
* Presence of clinical signs or symptoms of radiculopathy
* Diagnosis of spondylolisthesis
* Diagnosis of fibromyalgia
* Treatment with corticosteroids or other drugs in the previous two weeks
* History of spinal surgery
* Presence of central or peripheral system pathology (i.e. stroke, peripheral nerve etc.)
* Have received a physiotherapy treatment for low back pain before 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index(ODI) | Change between baseline and 4 weeks
  The Oswestry Disability Index(ODI) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. Scores between 0-5 are given for each question on the scale consisting of 10 questions. Questions are on travel, social life, sex life, sleeping, standing, sitting, walking, lifting things and personal precautions. Maximum score is 50, minimum score is 0.
Visual Analogue Scale(VAS) | Change between baseline and 4 weeks
  The Visual Analog Scale (VAS) is a scale used to determine the intensity of pain experienced by individuals. It consists of a line approximately 10-15 cm long; the patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain the left side means no pain with 0 points, while the right side means 10 points the worst pain ever.
Tampa Scale for Kinesiophobia(TSK) | Change between baseline and 4 weeks
  The Tampa Scale of Kinesiophobiais (TSK) is 17 items a self-reporting questionnaire based on evaluation of fear of movement, fear of physical activity, and fear avoidance. It was first developed to distinguish between non-excessive fear and phobia in patients with chronic musculoskeletal pain, specifically the fear of movement in patients with chronic low back pain then widely used for different parts of the body. The questionnaire using 4 points to assess that are based on; the model of fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury.(1 = Strongly Disagree, 4 = Strongly Agree).The total score of the scale range from 17-68, where 17 means no kinesiophobia, 68 means severe kinesiophobia.
Short Form(SF-36) | Change between baseline and 4 weeks
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It comprises 36 questions which cover eight domains of health:1) Limitations in physical activities because of health problems 2) Limitations in social activities because of physical or emotional problems 3) Limitations in usual role activities because of physical health problems 4) Bodily pain 5) General mental health (psychological distress and well-being) 6) Limitations in usual role activities because of emotional problems 7) Vitality (energy and fatigue) 8) General health perceptions. The SF-36 is often used as a measure of a person or population's quality of life (QOL). In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla ATAŞ BALCI, Assist Prof, Study Director — Bahçeşehir University
Locations (1):
- Private Medigold Sultan Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No